CLINICAL TRIAL: NCT04952805
Title: Randomized, Placebo-controlled, Double-blind, Multicenter, Seamless Adaptive Phase II-III Clinical Trial to Select the Dose and Evaluate Safety and Efficacy of MAD0004J08 Monoclonal Antibody in Adult Patients With Recently Diagnosed Asymptomatic to Moderately Severe COVID-19
Brief Title: Study to Select the Dose and Evaluate Safety and Efficacy of Monoclonal Antibody in Adult With Recently Diagnosed Asymptomatic to Moderately Severe COVID-19.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Toscana Life Sciences Sviluppo s.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0001B
Record Dates: First submitted 2021-07-01; First posted 2021-07-07 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — MAD0004J08

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Interventional Arm _400 mg (Experimental): To all the patients enrolled is admistrated with single dose of MAD0004J08 400 mg.
  Interventions: Drug: MAD0004J08
- Interventional Arm _100 mg (Experimental): To all the patients enrolled is admistrated with single dose of MAD0004J08 100 mg.
  Interventions: Drug: MAD0004J08
- Placebo Arm (Placebo Comparator): To all the patients enrolled is admistrated with single dose of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MAD0004J08 — MAD0004J08 is a human monoclonal Antibody (mAb), 2.5 mL 2R vial available in two dose: 100 mg and 400 mg. The pharmaceutical form is solution for intramuscular injection.
  Arms: Interventional Arm _100 mg; Interventional Arm _400 mg
Other: Placebo — Placebo matching to MAD0004J08, 2.5 mL 2R vial. The pharmaceutical form is solution for intramuscular injection.
  Arms: Placebo Arm

SUMMARY:
MAD0004J08, the experimental drug, is a potent neutralizing IgG1 monoclonal antibody (mAb) targeting the spike protein of SARS-CoV-2. MAD0004J08 blocks viral attachment and entry into human cells and neutralizes the virus. Because of its high affinity and potency, MAD0004J08 may accelerate clearance of the virus and prevent clinical deterioration of COVID-19 patients, especially when administered shortly after infection, and prevent SARS-CoV-2 infection in uninfected subjects. Because of its high potency, MAD0004J08 is expected to be effective at low doses (mg range) and thus will be administered by intramuscular (IM) injection, as opposed to the intravenous bolus required by high dose mAbs.

The goals of this Phase II-III seamless adaptive clinical trial are:

Stage-1 (Phase II)

1. Select one dose level for progression to Stage-2 Stage-1 + Stage-2 (Phase III)
2. Provide confirmatory evidence of safety and efficacy for regulatory approval.

DETAILED DESCRIPTION:
This clinical trial is designed as a randomized, stratified, placebo-controlled doubleblind, multicenter, seamless adaptive study. The target study population is adult patients ≥ 18 years of age with recently diagnosed (≤ 3 days from 1st positive swab taken) asymptomatic to moderately severe COVID-19 at baseline. Patients with comorbidities will be allowed in the study assuming all inclusion and exclusion criteria are met. Participants will not require hospitalization at baseline.

The trial is designed in two stages:

* Stage I: participants will be randomized (1:1:1 ratio) to one of the one of the following three study cohorts:
* MAD0004J08 400 mg, single dose
* MAD0004J08 100 mg, single dose
* Placebo, single dose The collected data will be analysed following a pre-planned interim analysis plan. Based on the results of this analysis the Data Monitoring Committee (DMC) will recommend whether the study should advance to Stage-2, and if so, will recommend selection of one of the two MAD0004J08 treatments for Stage-2. Alternatively, the DMC will recommend stopping the study. Final decisions will be made by an unblinded sub-group of the Steering Committee (SC), including senior Sponsor representatives, based on summary results.
* Stage-2: participants will be randomized (1:1 ratio) to one of two treatments:
* MAD0004J08, dose level selected in Stage-1, single dose
* Placebo, single dose Twelve (12) study visits and 2 telephone calls are scheduled for each participant over approximately 168 days. Additional ad-hoc visit(s) may be necessary to confirm eradication of SARS-CoV-2 from the upper respiratory tract (URT) following the 1st negative swab.

At Visit 1 (baseline) all participants will undergo testing for serum IgA and IgG vs. the spike (S) protein, and IgG vs. nucleocapsid (N) protein: participants testing negative to all three antibodies at baseline are referred to as seronegative; participants testing positive to any of the three antibodies at baseline are referred to as seropositive. Due to the need to minimize time between diagnosis and intervention, screening procedures, baseline procedures, randomization and administration of study treatment will occur on day 1.

Visits from Day 3 to Day 21 (Visits 2 to 9) will be conducted by study staff at the participant's home, unless the participant is hospitalized. Visits from Day 28 to Day 168 (Visits 10 to 12) will be conducted at the study center. Participants requiring hospitalization during the study period are to be hospitalized at the study center where Visit 1 was conducted.

At each scheduled visit nasopharyngeal swabs will be carried out. Additional swabs may be taken ad hoc to confirm eradication after the 1st negative swab.

Safety and efficacy endpoints will be analyzed as appropriate in two target populations (all randomized participants (ALL) and seronegative randomized participants (SEROneg) and three time-windows ( baseline (Visit 1) to end of Stage-1 or dropout (interim analysis), baseline (Visit 1) to end of Stage-2 or dropout (primary analysis) and baseline (Visit 1) to end of study (Visit 12) or dropout (final analysis).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent taken before any study procedure from any patient capable of giving consent, or, when the patient is incapable of doing so, by his or her legal/authorized representative.
* Age ≥18 years. At least 30% of participants will be ≥ 65 years old.
* First nasopharyngeal swab testing positive for SARS-CoV-2 by RT-PCR taken no more than 3 days before randomization (Visit 1). Results of "rapid" semiquantitative tests are not acceptable.
* Asymptomatic to moderately symptomatic outpatients with no need for immediate hospitalization: grade 1, or grade 2 or grade 3 of Clinical Severity Scale.
* No childbearing potential (post-menopause, surgically-induced, or pharmacologically-induced sterility) or, if of childbearing potential, negative urinary pregnancy test (women) and commitment to use at least 2 forms of contraception for at least 168 days from administration of study drug (men and women).

Exclusion Criteria:

* Severe or critical COVID-19: grade 4 or grade 5 of clinical severity scale.
* Current hospitalization and/or hospitalization or emergency room visit in the past 14 days.
* Need for immediate hospitalization for any reason in the investigator's opinion.
* Severe liver disease as determined by values of ALT and/or AST >5x upper limit of normal (ULN) and/or history of liver cirrhosis.
* Severe renal disease as determined by estimated creatinine clearance (CcCl) <30 mL/min or serum creatinine >2 mg/dL (>176.8 μmol/L) or ongoing renal dialysis.
* Absolute neutrophil count (ANC) < 1000/μL.
* Demyelinating and connective tissue disease.
* Active tuberculosis or suspected active bacterial, fungal, viral, or other infection (besides COVID- 19).
* Any condition that in the Investigator's opinion may be negatively affected by the study treatments and/or study procedures.
* Any condition, including psychiatric disorders, alcohol, or substance abuse, which in the Investigator's opinion may interfere with completion of the study procedures.
* Any condition with life expectancy <6 months in the Investigator's opinion.
* Ongoing or planned pregnancy.
* Ongoing breast feeding.
* History of life-threatening event in the 1 month before Visit 1.
* History of surgery in the 1 month before Visit 1.
* History of treatment with blood components in the 6 months before Visit 1.
* History of cancer treated with chemotherapy in the 6 months before Visit 1.
* History of solid organ transplant at any time before Visit 1.
* History of severe and/or serious allergic reaction to monoclonal antibodies or any component of MAD0004J08, including anaphylaxis at any time before Visit 1.
* Treatment with an investigational drug or vaccine within 5 half-lives or 30 days (whichever is longer) of randomization.
* Treatment at any time with monoclonal antibodies bamlanivimab, bamlanivimab + etesevimab combination, and casiribimab + imdevimab combination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2021-06-06 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Severe (Grade 3) unsolicited AEs and/or serious unsolicited AEs (SAEs). | From admission to discharge - Assessed as day 0
  Proportion of participants with severe (Grade 3) unsolicited AEs and/or serious unsolicited AEs (SAEs).
Time to SARS-CoV-2 clearance in the URT. | From baseline (visit 1) up to day 168 ± 7 (visit 12)
  Evaluation of the time required for the elimination of SARS-CoV-2 in the URT.

SECONDARY OUTCOMES:
Unsolicited AEs, including clinically relevant laboratory and ECG abnormalities. | From baseline (visit 1) up to day 168 ± 7 (visit 12)
  Proportion of participants with unsolicited AEs, including clinically relevant laboratory and ECG abnormalities.
Solicited local AEs at the injection site | From baseline (visit 1) up to day 28 (Visit 10)
  Proportion of participants with solicited local AEs at the injection site. Will be considered: pain, swelling and redness at the injection site.
Number of participants who develop ADA. | At baseline (visit 1), at day 7 (visit 4), at day 28 (visit 10), at day 56 ± 7 (visit 11) and at day 168 ± 7 (visit 12)
  Proportion of participants who develop ADA. The first 60 randomized participants will be tested for ADA.
SARS-CoV-2 clearance in the URT | At baseline (visit 1), at day 7 (visit 4), at day 28 (visit 10), at day 56 ± 7 (visit 11) and at day 168 ± 7 (visit 12)
  Proportion of participants with SARS-CoV-2 clearance in the Upper Respiratory Tract (URT) at each visit.
SARS-CoV-2 viral load in nasopharyngeal swab | From baseline (visit 1) up to day 168 ± 7 (visit 12)
  SARS-CoV-2 viral load (number of copies) in nasopharyngeal swab, as measured by RT-PCR at each visit.
SPO2% and lowest SpO2 % post baseline. | From baseline (visit 1) up to day 168 ± 7 (visit 12)
  SPO2 % value at each visit and lower SpO2 % after baseline.
SpO2 % < 94%. | From baseline (visit 1) up to day 168 ± 7 (visit 12)
  Proportion of participants with SpO2 % < 94%.
Participants with increased dose home oxygen therapy | From baseline (visit 1) up to day 168 ± 7 (visit 12)
  Proportion of participants with newly established or increased dose home oxygen therapy increased home oxygen therapy (only applies to patients with underlying conditions other than COVID-19 requiring such therapy, e.g., COPD).
Area under the curve (AUC) of COVID-19 total symptom score (range: 0-24). | From baseline (visit 1) up to day 168 ± 7 (visit 12)
  Assessment of COVID-19 total symptom score
Participants requiring hospitalization | From event start (day 0) through event completion
  Proportion of participants requiring hospitalization.
Cumulative time of hospital stay in days. | From event start (day 0) through event completion
  Number of days the participant was hospitalised
Hospitalized participants requiring supplemental oxygen therapy. | From event start (day 0) through event completion
  Proportion of hospitalized participants requiring supplemental oxygen therapy.
Cumulative time of hospitalized oxygen therapy in days. | From event start (day 0) through event completion
  Number of days the hospitalized participant required oxygen therapy
Participants admitted to intensive care unit (ICU). | From event start (day 0) through event completion
  Proportion of participants admitted to intensive care unit (ICU).
Cumulative time of ICU stay in days. | From event start (day 0) through event completion
  Number of days the hospitalized participant stay in therapy intensive care unit
All-cause mortality. | From baseline (visit 1) to through study completion
  Analysis of all All-cause mortality.
MAD0004J08 serum concentration. | From baseline (visit 1) up to day 168 ± 7 (visit 12)
  Evaluation of MAD0004J08 serum concetration

CONTACTS AND LOCATIONS:
Overall Officials: Simone Lanini, Principal Investigator — IRCCS INMI Lazzaro Spallanzani - Istituto nazionale Malattie Infettive
Locations (14):
- Italy (14):
  - IRCCS INMI Lazzaro Spallanzani - Istituto nazionale Malattie Infettive, Roma, RM
  - Az. Ospedaliera San Giuseppe Moscati, Avellino
  - Azienda Ospedaliero-Universitaria Careggi di Firenze, Florence
  - A.O. Ospedali Riuniti di Foggia - Università degli Studi di Fog, Foggia
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan
  - Az. Ospedaliera dei Colli - P.O. "D. Cotugno", Napoli
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia
  - Azienda USL Ospedale "Guglielmo da Saliceto", Piacenza
  - A.O.U. Pisana - Ospedale di Cisanello, Pisa
  - Policlinico Santa Maria alle Scotte - Università di Siena, Siena
  - Ospedale di Cattinara, Trieste
  - ASL di Vercelli - Ospedale Sant'Andrea, Vercelli
  - A.O.U. Integrata di Verona, Verona

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343